CLINICAL TRIAL: NCT03018964
Title: A Prospective Multicenter Randomized Controlled Study for The Safety of Single Incision Laparoscopic Cholecystectomy With a Camera Holder Versus With a Camera Operator
Brief Title: Solo Single Incision Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Chungbuk National University Hospital (Other); Gyeongsang National University Hospital (Other)
Responsible Party: Principal Investigator, YoungRok Choi, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SILC_HoOp
Record Dates: First submitted 2017-01-08; First posted 2017-01-12 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Cholecystectomy, Laparoscopic
Keywords: Single incision; Solo surgery
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solo-SILC (Experimental): Solo surgery using a laparoscopic camera holder instead of a camera operator in SILC
  Interventions: Procedure: Solo surgery
- Ca-SILC (Active Comparator): No solo surgery, operation with a camera operator in SILC
  Interventions: Procedure: operation with a camera operator in SILC

INTERVENTIONS:
Procedure: Solo surgery — Solo surgery using a camera scope holder in single incision laparoscopic cholecystectomy
  Arms: Solo-SILC
Procedure: operation with a camera operator in SILC — conventional single incision laparoscopic cholecystectomy with a scopist
  Arms: Ca-SILC

SUMMARY:
The purpose of this study is to determine safety of solo surgery in single incision laparoscopic cholecystectomy (SILC) with a camera holder comparing to a camera operator assisted SILC

DETAILED DESCRIPTION:
This study is a multicenter randomized controlled study. The primary outcome based on non-inferior study design(α=0.05, power (1-β)=0.90); comparing a complications rate between Solo-SILC group and conventional cholecystectomy group (Ca-SILC).

Total of 272 patients who were undergoing laparoscopic cholecystectomy for gallbladder disorders will randomly assign to two groups according to a computer-generated table of random numbers Solo-SILC group using a laparoscopic camera holder (n=136) or Ca-SILC group in which a camera operator joins (n=136). .

Demographics (i.e., age, gender, body mass index (BMI), American Society of Anesthesiology (ASA) score, indication for operation, need for conversion to open surgery or additional port will be recorded. Outcome including pain, hernia, complication rates, post-cholecystectomy diarrhea, operator's workload will be investigated

ELIGIBILITY:
Inclusion Criteria:

* all patient need laparoscopic cholecystectomy (check the possibility of routine application of Solo-SILC in clinical practice)

Exclusion Criteria:

* Mirizzi syndrome
* unstable vital sign
* no compliance
* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Complication rate in Solo-Single Incision Laparoscopic Cholecystectomy (SILC) | average 2 weeks
  intraoperative and immediate postoperative complications in Solo-SILC comparing with that in laparoscopic cholecystectomy

SECONDARY OUTCOMES:
complications in both groups | average 2 weeks
  intraoperative and postoperative complications
Conversion rate | intraoperative
  intraoperative conversion rate to open or additional port surgery
Incisional hernia | average 6 months
  Umbilical incisional hernia incidence
Wound, back, and shoulder pain | postoperative 6 hr, 24 hr, 2 weeks after the operation
  Access the patient's pain using the visual analog scale
Postoperative adverse symptoms after SILC | average 2weeks after discharge
  Diet change, post-cholecystectomy diarrhea
number of participant with abnormal laboratory values | average 2weeks after discharge
  postoperative laboratory findings on visiting outpatient's clinic
Operator's workload | intraoperative
  Access a operator's workload just after solo surgery comparing to Ca-SILC group using NASA Task Load Index (NASA-TLX) score

CONTACTS AND LOCATIONS:
Overall Officials: Soyeon Ahn, Ph.D., Principal Investigator — Medical Research Collaboration Center Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Navarra G, Pozza E, Occhionorelli S, Carcoforo P, Donini I. One-wound laparoscopic cholecystectomy. Br J Surg. 1997 May;84(5):695. No abstract available. PMID 9171771
- [Result] Tsimoyiannis EC, Tsimogiannis KE, Pappas-Gogos G, Farantos C, Benetatos N, Mavridou P, Manataki A. Different pain scores in single transumbilical incision laparoscopic cholecystectomy versus classic laparoscopic cholecystectomy: a randomized controlled trial. Surg Endosc. 2010 Aug;24(8):1842-8. doi: 10.1007/s00464-010-0887-3. Epub 2010 Feb 20. PMID 20174950
- [Result] Marks J, Tacchino R, Roberts K, Onders R, Denoto G, Paraskeva P, Rivas H, Soper N, Rosemurgy A, Shah S. Prospective randomized controlled trial of traditional laparoscopic cholecystectomy versus single-incision laparoscopic cholecystectomy: report of preliminary data. Am J Surg. 2011 Mar;201(3):369-72; discussion 372-3. doi: 10.1016/j.amjsurg.2010.09.012. PMID 21367381
- [Result] Markar SR, Karthikesalingam A, Thrumurthy S, Muirhead L, Kinross J, Paraskeva P. Single-incision laparoscopic surgery (SILS) vs. conventional multiport cholecystectomy: systematic review and meta-analysis. Surg Endosc. 2012 May;26(5):1205-13. doi: 10.1007/s00464-011-2051-0. Epub 2011 Dec 16. PMID 22173546
- [Result] Phillips MS, Marks JM, Roberts K, Tacchino R, Onders R, DeNoto G, Rivas H, Islam A, Soper N, Gecelter G, Rubach E, Paraskeva P, Shah S. Intermediate results of a prospective randomized controlled trial of traditional four-port laparoscopic cholecystectomy versus single-incision laparoscopic cholecystectomy. Surg Endosc. 2012 May;26(5):1296-303. doi: 10.1007/s00464-011-2028-z. Epub 2011 Nov 15. PMID 22083331
- [Result] Deveci U, Barbaros U, Kapakli MS, Manukyan MN, Simsek S, Kebudi A, Mercan S. The comparison of single incision laparoscopic cholecystectomy and three port laparoscopic cholecystectomy: prospective randomized study. J Korean Surg Soc. 2013 Dec;85(6):275-82. doi: 10.4174/jkss.2013.85.6.275. Epub 2013 Nov 26. PMID 24368985
- [Result] Gillen S, Pletzer B, Heiligensetzer A, Wolf P, Kleeff J, Feussner H, Furst A. Solo-surgical laparoscopic cholecystectomy with a joystick-guided camera device: a case-control study. Surg Endosc. 2014 Jan;28(1):164-70. doi: 10.1007/s00464-013-3142-x. Epub 2013 Aug 29. PMID 23990155
- [Result] Sasaki K, Watanabe G, Matsuda M, Hashimoto M. Original single-incision laparoscopic cholecystectomy for acute inflammation of the gallbladder. World J Gastroenterol. 2012 Mar 7;18(9):944-51. doi: 10.3748/wjg.v18.i9.944. PMID 22408354
- [Result] Chuang SH, Chen PH, Chang CM, Lin CS. Single-incision vs three-incision laparoscopic cholecystectomy for complicated and uncomplicated acute cholecystitis. World J Gastroenterol. 2013 Nov 21;19(43):7743-50. doi: 10.3748/wjg.v19.i43.7743. PMID 24282363
- [Result] Sinha R, Yadav AS. Transumbilical single incision laparoscopic cholecystectomy with conventional instruments: A continuing study. J Minim Access Surg. 2014 Oct;10(4):175-9. doi: 10.4103/0972-9941.141502. PMID 25336816
- [Result] Saber AA, El-Ghazaly TH, Dewoolkar AV, Slayton SA. Single-incision laparoscopic sleeve gastrectomy versus conventional multiport laparoscopic sleeve gastrectomy: technical considerations and strategic modifications. Surg Obes Relat Dis. 2010 Nov-Dec;6(6):658-64. doi: 10.1016/j.soard.2010.03.004. Epub 2010 Mar 19. PMID 20727831
- [Result] Strasberg SM, Hertl M, Soper NJ. An analysis of the problem of biliary injury during laparoscopic cholecystectomy. J Am Coll Surg. 1995 Jan;180(1):101-25. No abstract available. PMID 8000648